CLINICAL TRIAL: NCT04427267
Title: Assessment of Thermal Condition of Health Workers Who Use Personal Protective Equipment for Biological Factors During Their Work With COVID-19 Patients
Brief Title: Assessment of Thermal Condition of Health Workers Who Use Personal Protective Equipment From Biological Hazards During Their Work With COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Federal State Budgetary Scientific Institution "Izmerov Research Institute of Occupational Health" (Other)
Responsible Party: Principal Investigator, Andrey Mikhailovich Geregey, Head of the Laboratory of Personal Protective Equipment and Industrial Exoskeletons Andrey Geregey, Federal State Budgetary Scientific Institution "Izmerov Research Institute of Occupational Health"
Other Study IDs: PPE-02
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Thermal Condition of Health Workers Who Use Personal Protective Equipment From Biological Hazards During Their Work With COVID-19 Patients
Keywords: Thermophysiology; Personal protective equipment from biological hazards; Medical workers; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health workers
  Interventions: Other: Personal protective equipment from biological hazard

INTERVENTIONS:
Other: Personal protective equipment from biological hazard — Includes: isolation clothing, mask, eyewear, overshoes

SUMMARY:
This research will provide data on thermal condition of medical workers who use personal protective equipment from biological hazards. Aquired data will be used to define acceptable period of use for these protective costumes.

This research will recruit 6 volunteers. During 6 hours each subject will perform their work using protective costume. Heart rate, skin and air temperature under costume and hygrometric data will be registered. Also there will be questionnaires for volunteers for subjective assessment of thermal and moisture sensations.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals (based on medical screening)

Exclusion Criteria:

* endocrinological diseases and disorders
* health deviations at the time of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Health workers
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-06-27 (Actual); Study Completion 2020-06-27 (Actual)

PRIMARY OUTCOMES:
Skin thermometry | 6 hours
  DS1923-F5 Thermochron iButtons
Hygrometry under costume | 6 hours
  DS1923-F5 Thermochron iButtons
Heart rate | 6 hours
  A Polar H10 heart rate monitor (Polar Electro, Finland) will carry all items during the entire research
Air thermometry | 6 hours
  Meteoscop - M
Air hygrometry | 6 hours
  Meteoscop - M

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Scientific Institution Izmerov Research Institute of Occupational Health, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No